CLINICAL TRIAL: NCT03028896
Title: Comparison of Standard Versus 90° Rotation Technique for LMA FlexibleTM Insertion
Brief Title: 90° Rotation Technique for LMA FlexibleTM Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, associator professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SNU-LMA
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Laryngeal Masks
Keywords: LMA Flexible

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard (No Intervention): In the neck flexed and the head extended position, hold mask like a pen with the index finger placed anteriorly at the junction of the cuff and tube, push the mask backwards maintaining pressure against the palate until resistance is felt.
- rotational (Experimental): After insertion of the entire cuff inside the mouth, the LMA FlexibleTM was rotated counter-clockwise through 90° and was advanced through the right side of the tongue until the resistance was felt, and then was returned back in the hypopharynx.
  Interventions: Procedure: 90° rotational technique

INTERVENTIONS:
Procedure: 90° rotational technique — the LMA FlexibleTM was rotated counter-clockwise through 90°
  Arms: rotational

SUMMARY:
The 90° rotation technique is known to improve the success rate of conventional LMA but its effect in LMA FlexibleTM is not known. We tried to find if 90° rotation technique could increase the first attempt success rate of the insertion of LMA FlexibleTM compared to standard technique.

DETAILED DESCRIPTION:
One hundred and sixteen adult patients undergoing breast surgery were randomized to the two insertion techniques. The ease of insertion was assessed by the success rate at the first attempt. Heart rate and mean blood pressure were recorded 1 min before and 1 min after insertion. Postoperative complications were checked.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I - II
* Scheduled for elective breast surgery under general anaesthesia using LMA FlexibleTM

Exclusion Criteria:

* known difficult airway
* mouth opening less than 2.5 cm
* limited extension of neck
* recent sore throat
* gastroesophageal reflux disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast surgery
Enrollment: 132 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2017-01-19 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Koo BW, Oh AY, Hwang JW, Na HS, Min SW. Comparison of standard versus 90 degrees rotation technique for LMA Flexible insertion: a randomized controlled trial. BMC Anesthesiol. 2019 Jun 7;19(1):95. doi: 10.1186/s12871-019-0773-z. PMID 31170926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard | Rotational
Started | 66 | 66
Completed | 63 | 66
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Rotational | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 62 | 62 | 124
  >=65 years | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 129
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate
Description: the first attempt success rate of insertion of LMA FlexibleTM
Time Frame: at induction
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Rotational
Number analyzed (Participants) | 63 | 66
Participants | 59 | 65

2. Secondary Outcome: Insertion Time
Description: time from passed mouth of the device to the effective ventilation after inflation of the cuff
Time Frame: at induction
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Standard | Rotational
Number analyzed (Participants) | 63 | 66
seconds | 10.5 (4.7) | 9.7 (4.7)

3. Secondary Outcome: Oropharyngeal Leak Pressure
Description: audible leak during manual ventilation at mouth
Time Frame: at induction
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Standard | Rotational
Number analyzed (Participants) | 63 | 66
cmH2O | 19.8 (4.9) | 20.5 (4.2)

4. Secondary Outcome: Number of Participants With Blood Staining on the Laryngeal Mask Airway
Description: Number of Participants with blood staining on the laryngeal mask airway.
Time Frame: post op 1min
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Rotational
Number analyzed (Participants) | 63 | 66
Participants | 1 | 3

ADVERSE EVENTS:
Arm/Group | Standard | Rotational
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No